CLINICAL TRIAL: NCT02785887
Title: Impact of Geriatrician-implemented Interventions on Chemotherapy Delivery in Vulnerable Elderly Patients With Early or Metastatic Solid Malignancies: the GIVE Trial
Brief Title: Impact of Geriatrician Interventions on Chemotherapy Delivery in Vulnerable Elderly Oncology Patients
Acronym: GIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL 4 Prato (Other)
Responsible Party: Principal Investigator, Laura Biganzoli, MD, Azienda USL 4 Prato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GIVE
Record Dates: First submitted 2014-03-26; First posted 2016-05-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer; Bladder Cancer; Gastrointestinal Cancer
Keywords: Breast cancer; lung cancer; Gastrointestinal Cancer; Ovarian cancer; Prostate cancer; bladder cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oncological and geriatrician review (Experimental): Routine oncological care plus geriatric intervention
  Interventions: Other: Geriatrician review
- Oncological care (No Intervention): Routine oncological care only

INTERVENTIONS:
Other: Geriatrician review — In addition to routine oncological care, patients will be reviewed by a geriatrician and may receive intervention if CGA deficits are found
  Arms: Oncological and geriatrician review

SUMMARY:
This is a randomized parallel group trial designed to evaluate the impact of implementing geriatrician-prescribed interventions based on the comprehensive geriatric assessment (CGA), on the ability to deliver adequate chemotherapy treatment, as measured by relative dose intensity (RDI).

DETAILED DESCRIPTION:
This randomized parallel group trial is designed to evaluate the impact of implementing geriatrician-prescribed interventions, on the ability to deliver adequate chemotherapy treatment, as measured by RDI of at least 85%, in a cohort of vulnerable [≥1 deficit identified at CGA and/or ≥1 comorbidity Grade 3-4 as defined by Cumulative Illness Rating Scale for Geriatrics (CIRS-G)] elderly cancer patients with early stage or advanced solid organ malignancies.

Patients will be randomized using a 2:1 allocation to Arm A: routine oncological care plus geriatric intervention or Arm B: routine oncological care

ELIGIBILITY:
Inclusion Criteria:

1. Any solid tumors
2. Either early stage disease planned for treatment with neo/adjuvant chemotherapy, or metastatic disease planned for treatment with chemotherapy and ≤ 1 previous chemotherapy treatment in the metastatic setting
3. Absence of symptomatic central nervous system (CNS) metastases
4. Eastern Cooperative Oncology group (ECOG) performance status 0-2
5. Estimated life expectancy of ≥ 12 weeks
6. At least 1 deficit identified on CGA at screening/baseline, and/or at least one comorbidity of grade 3 or 4 severity, as defined by CIRS-G
7. Written informed consent in according to International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use/Good Clinical Practice (ICH/GCP), and national/local ethics regulations
8. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up schedule

Exclusion Criteria:

1. Age ≤ 69 years
2. Any patients who did not meet the inclusion criteria

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 233 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Relative dose intensity | 6 months
  Relative dose intensity (RDI) is defined as the ratio (in percentage) of the total administered dose of chemotherapy to the standard dose of the same chemotherapy regimen, as defined by the treating centre. RDI will be calculated as the total dose delivered from the first day of cycle 1 of chemotherapy until completion of the planned chemotherapy (average of 6 months for early, 3 months for metastatic disease), or until date of relapse or death or discontinuation from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Occurrence of treatment-related toxicity | every 3-4 weeks up to 6 months
  Severity will be reported based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Occurrence of hospitalization | at 6 months for early and at 3 months for metastatic disease
  Documentation of hospitalization
Early mortality | death from any cause occurring 12 months of randomization for neo/adjuvant patients, or within 6 months for patients with metastatic disease
  Documentation of death

OTHER OUTCOMES:
Optional Translational Substudy: Blood metabolites | up to 12 months
  Proton Nuclear Magnetic Resonance (H-NMR) metabolomics spectra will be derived from a 10ml fasting peripheral serum sample collected prior to commencing chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Laura Biganzoli, MD, Principal Investigator — Azienda USL 4 Prato
Locations (3):
- Italy (3):
  - Ospedale Vito Fazi, Lecce
  - Ospedale San Paolo, Milan
  - Istituto Oncologico Veneto, Padua

IPD SHARING:
Plan to Share IPD: No